CLINICAL TRIAL: NCT02721355
Title: Evaluation of a Health Food Supplement Containing Anti-Helicobacter Pylori Urease IgY Antibody on Patients With Chronic Gastritis in Hanoi, Vietnam
Brief Title: Effect of Chicken Egg Antibody (IgY) on Patients With Chronic Gastritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Immunology Research Institute in Gifu (Industry)
Collaborators: Dong Do Pharmaceutical Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BV108-15
Record Dates: First submitted 2016-03-03; First posted 2016-03-29 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2016-08

CONDITIONS: Chronic Gastritis Caused by Helicobacter Pylori
Keywords: Chronic gastritis; Gastric ulcer; Helicobacter pylori; IgY
MeSH Terms: conditions — Stomach Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Food supplement GastimunHP (Experimental): The subjects take food supplement containing specific IgY (GastimunHP) during treatment with routine medical regime
  Interventions: Dietary Supplement: GastimunHP
- Control (No Intervention): The subjects undergo the routine treatment regime without taking food supplement

INTERVENTIONS:
Dietary Supplement: GastimunHP — Health food supplement containing specific IgY against urease of H. pylori
  Arms: Food supplement GastimunHP

SUMMARY:
H. pylori positive patient volunteers that passed the selection criteria are recruited and divided into a test and a control group. Both groups are treated with a current treatment regime (EAC: Esomeprazole 40 mg/day; Clarithromycin 1000 mg/day; Amoxicillin 2000 mg/day) but only the test group received IgY-containing food supplement as an adjunctive measure for 15 days. The subjects are examined before and 4 weeks after the treatment initiation by Urea Breath Test (UBT) and gastro-endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastritis or gastric ulcer who are positive to H. pylori

Exclusion Criteria:

* People allergic to egg proteins

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-06; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khien V Vu, Ph. D, Principal Investigator — Dept. of Diagnostic Endoscopy, 108 Military Central Hospital, Hanoi, Vietnam
Locations (1):
- 108 Military Central Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Food Supplement GastimunHP | Control
Started | 42 | 42
Completed | 36 | 41
Not Completed | 6 | 1
Not completed — Lost to Follow-up | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Food Supplement GastimunHP | Control | Total
Number analyzed (Participants) | 36 | 41 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (12.7) | 44.2 (12.5) | 46.05 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 22 | 38
  Male | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: UBT Values at Baseline and 8 Weeks
Description: Urea Breath test (UBT) value was examined at baseline (0 week) and 8 weeks later. A commercial kit was used following the instructions from the manufacturer. A cut off value of 50 is considered to be positive. Higher UBT values indicate worse outcome.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: UBT value
Arm/Group | Food Supplement GastimunHP | Control
Number analyzed (Participants) | 36 | 41
UBT value
  Baseline | 161.64 (83.53) | 158.54 (43.73)
  After 8 weeks | 49.42 (44.21) | 73.37 (30)

2. Secondary Outcome: Number of Participants With a Reduction in Severity of Abdominal Pain at 1 and 4 Weeks
Description: Outcome measures are the Gastrointestinal Symptom Rating Scale (GSRS) scores using a four-point graded scale (0 = none: no symptoms; 1 = mild: awareness of sign or symptom, but easily tolerated; 2 = moderate: discomfort sufficient to cause interference with normal activities; 3 = severe: incapacitating with inability to perform normal activities).
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Food Supplement GastimunHP | Control
Number analyzed (Participants) | 36 | 41
Participants
  Reduced pain after 1 week | 19 | 16
  Reduced pain after 4 weeks | 25 | 25

3. Secondary Outcome: Number of Participants With a Reduction in Gastrointestinal Symptom Rating Scale (GSRS) Scores at 1 and 4 Weeks
Description: Outcome measures are the Gastrointestinal Symptom Rating Scale (GSRS) scores using a four-point graded scale (0 = no nausea; 1 = occasional episodes of short duration; 2 = frequent and prolonged nausea, no vomiting; 3 = continuous nausea, frequent vomiting)
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Food Supplement GastimunHP | Control
Number analyzed (Participants) | 36 | 41
Participants
  Number of participants with reduced GSRS scores after 1 week | 18 | 15
  Number of participants with reduced GSRS scores after 4 weeks | 25 | 25

4. Other Pre Specified Outcome: Number of Participants With Reduced Bloating After 1 Week
Description: Participants were asked to monitor stomach bloating after each meal daily during the first week of treatment. The participants that felt having less bloating were recorded to have reduced bloating.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Food Supplement GastimunHP | Control
Number analyzed (Participants) | 36 | 41
Participants | 18 | 15

ADVERSE EVENTS:
Arm/Group | Food Supplement GastimunHP | Control
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/41
Other Adverse Events (participants affected / at risk) | 1/36 | 0/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Food Supplement GastimunHP (N=36) | Control (N=41)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No